CLINICAL TRIAL: NCT04900558
Title: Impact of Robotic Surgery on Post-operative Outcomes of Patients Who Underwent Radical Cystectomy
Brief Title: Robotic Radical Cystectomy Outcomes
Status: Recruiting | Type: Observational
Sponsor: University of Florence (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Simone Morselli, PhD Student, University of Florence
Other Study IDs: 19303_oss
Record Dates: First submitted 2021-05-03; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Bladder Cancer; Muscle-Invasive Bladder Carcinoma; Oncology; Recurrence; Surgery
Keywords: Cystectomy; Radical Cystectomy; Ileal Conduit; Neobladder; Bladder Cancer; Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasms; Recurrence | interventions — Cystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Radical Cystectomy: Patients who underwent radical cystectomy for bladder cancer in our centre
  Interventions: Procedure: Radical Cystectomy

INTERVENTIONS:
Procedure: Radical Cystectomy — All the patients enrolled have undergone or will undergo radical cystectomy, with or without lymphadenectomy or urethrectomy All possibles urinary diversion are included, like ileal conduit, neobladder etc...

SUMMARY:
Currently, in the treatment of bladder cancer the use of robotics has entered in clinical practice, therefor robotic radical cystectomy with or without reconstruction is offered to patients during counseling procedures, if deemed appropriate and possible. The aim of the study is therefore the long-term evaluation of the peri-post-operative, oncological and functional results of patients undergoing radical cystectomy, both with an open and robotic approach. This study will thus help to clarify the actual impact of robotic surgery

ELIGIBILITY:
Inclusion Criteria:

* Age major or equal 18 years
* Patients who will undergo radical cystectomy
* Consent to participate

Exclusion Criteria:

* Absence of willingness to participate
* Further refusal to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is made up of patients who underwent radical cystectomy at AOU Careggi, SOD Robotic Urological Surgery, Minimally Invasive and Renal Transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2031-02-01 (Estimated); Study Completion 2038-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who will die from bladder cancer | From enrollment to late follow-up, up to 7 years
  Bladder Cancer Specific Mortality after surgery
Number of participants who will experience bladder cancer recurrence | From enrollment to late follow-up, up to 7 years
  Bladder Cancer Recurrence
Number of participants who will die from all causes | From enrollment to late follow-up, up to 7 years
  All cause mortality after surgery

SECONDARY OUTCOMES:
Number of participants who will die from bladder cancer after Robotic Surgery | From enrollment to late follow-up, up to 7 years
  Robotic surgery specific impact on survival
Number of participants who will experience bladder cancer recurrence after Robotic Surgery | From enrollment to late follow-up, up to 7 years
  Robotic surgery specific impact on recurrence
Number of participants who will experience surgical complications after Robotic Surgery | From enrollment to late follow-up, up to 7 years
  Robotic surgery specific impact on surgical complications
Variation in Quality of Life questionnaire after Robotic Surgery | From enrollment to late follow-up, up to 7 years
  Robotic surgery specific impact on quality of life according to European Organisation for Research and Treatment of Cancer (EORTC) core quality of life questionnaire (QLQ-C30)
Variation in Quality of Life questionnaire according to Urinary diversions | From enrollment to late follow-up, up to 7 years
  Urinary diversion specific impact on quality of life according to European Organisation for Research and Treatment of Cancer (EORTC) core quality of life questionnaire (QLQ-C30)
Number of participants who will experience surgical complications according to Urinary diversions | From enrollment to late follow-up, up to 7 years
  Urinary diversion specific impact on surgical complications
Number of participants who will experience bladder cancer recurrence according to Urinary diversions | From enrollment to late follow-up, up to 7 years
  Urinary diversion specific impact on bladder cancer recurrence
Number of participants who will die from bladder cancer according to Urinary diversions | From enrollment to late follow-up, up to 7 years
  Urinary diversion specific impact on bladder cancer rmortality
Number of participants who will die from all causes according to Urinary diversions | From enrollment to late follow-up, up to 7 years
  Urinary diversion specific impact on all cause mortality after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Arcangelo Sebastianelli, MD, Principal Investigator — Careggi Hospital, University of Florence; Sergio Serni, Prof, Principal Investigator — University of Florence; Simone Morselli, MD, Principal Investigator — University of Florence
Locations (1):
- Careggi University Hospital, Florence, Tuscany, Italy